CLINICAL TRIAL: NCT06403371
Title: The Effect of Fluoride Varnish on White Spot Lesion in Clear Aligner Orthodontic Patients: Prospective Randomized Controlled Clinical Trial
Brief Title: The Effect of Fluoride Varnish on White Spot Lesion in Clear Aligner Orthodontic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Suzan Al-Khateeb, Professor in Orthodontics, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JUST20230273
Record Dates: First submitted 2024-04-16; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: White Spot Lesion
Keywords: Fluoride varnish; Clear aligners; White spot lesions; Quantitative light induced fluorescence (QLF)
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Nor the subjects neither the investigator knew the type of varnish they received. Additionally, the outcome assessor was blinded before making the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride varnish group (Experimental): Patients received a layer of fluoride varnish on their teeth before the start of orthodontic clear aligner therapy
  Interventions: Other: Fluoride varnsh
- Control group (Placebo Comparator): Patients received a layer of normal saline on their teeth before the start of orthodontic clear aligner therapy
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Fluoride varnsh — Fluoride varnish was applied to the teeth surfaces before aligner therapy
  Arms: Fluoride varnish group
Other: Normal saline — Normal saline was applied to the teeth surfaces before aligner therapy
  Arms: Control group

SUMMARY:
Fluoride varnish is being applied on the teeth surfaces of patients undergoing orthodontic treatment just before receiving their clear aligners. The effect of the varnish was investigated if it can reduce the incidence of enamel demineralization or not.

DETAILED DESCRIPTION:
Background: The preventive effect of fluoride varnish on the development of white spot lesions (WSLs) during clear aligner treatment has not been investigated in the literature. Hence this was the purpose of this study. Material and Methods: This was a prospective double-blinded randomized clinical trial. A total of 44 patients (7 males, 37 females, with a mean age of 20.91 ± 4.56) who sought clear aligner therapy at the postgraduate orthodontic clinics at JUST were recruited and randomly divided equally (n=22 in each group) by a website randomizer. Eligibility criteria included healthy patients of both sexes (age range 14-30 years), Class I malocclusion with mild-to-moderate crowding (≤5 mm), non-extraction treatment plan, and optimum oral hygiene before treatment. Both the patient and the investigator were blinded during the intervention and assessment of outcomes. At (T0) Fluoride varnish was applied to the subjects in Group 1, while normal saline was applied to the subjects in Group 2 as a control. Quantitative light-induced fluorescence (QLF) images were taken at the start of the treatment (T0) and after 4 months (T1). The QLF images were analyzed to assess the primary outcomes: lesion area (Pixels), the mean amount of fluorescence loss (ΔF)% in addition to the number of newly developed lesions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects form both sexes
* Mild to moderate crowding
* Optimum oral hygiene
* Maximum of three restored teeth

Exclusion Criteria:

* Presence of enamel hypoplasia or hypocalcification,
* Any salivary gland disease or medication use that affect the salivary flow
* Subjects using fluoride other than 1450 ppm fluoride toothpaste.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Average lesion fluorescence loss (∆F%) | 4 months
  It reflects amount of mineral loss
Maximum lesion fluorescence loss (∆F-max%) | 4 months
  It measures the deepest point of the lesion (in relation to sound enamel) using QLF system in percent
Lesion area | 4 months
  It measures white spot lesion area in pixels

SECONDARY OUTCOMES:
Plaque measurement | 4 months
  It measures the amount of plaque on teeth surfaces in percent using QLF system

CONTACTS AND LOCATIONS:
Overall Officials: Susan Al-Khateeb, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Postgraduate Teaching Clinics/JUST, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zabokova-Bilbilova E, Popovska L, Kapusevska B, Stefanovska E. White spot lesions: prevention and management during the orthodontic treatment. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2014;35(2):161-8. doi: 10.2478/prilozi-2014-0021. PMID 25532098
- [Background] Ogaard B. [Cariologic aspects of orthodontic treatment]. Nor Tannlaegeforen Tid. 1989 Dec;99(20):802-5. Norwegian. PMID 2640705
- [Background] Boersma JG, van der Veen MH, Lagerweij MD, Bokhout B, Prahl-Andersen B. Caries prevalence measured with QLF after treatment with fixed orthodontic appliances: influencing factors. Caries Res. 2005 Jan-Feb;39(1):41-7. doi: 10.1159/000081655. PMID 15591733
- [Background] Sharma S, Narkhede S, Sonawane S, Gangurde P. Evaluation of Patient's Personal Reasons and Experience with Orthodontic Treatment. J Int Oral Health. 2013 Dec;5(6):78-81. Epub 2013 Dec 26. PMID 24453449
- [Background] van der Veen MH, de Josselin de Jong E. Application of quantitative light-induced fluorescence for assessing early caries lesions. Monogr Oral Sci. 2000;17:144-62. doi: 10.1159/000061639. PMID 10949838
- [Background] Geiger AM, Gorelick L, Gwinnett AJ, Benson BJ. Reducing white spot lesions in orthodontic populations with fluoride rinsing. Am J Orthod Dentofacial Orthop. 1992 May;101(5):403-7. doi: 10.1016/0889-5406(92)70112-N. PMID 1590288
- [Background] Rossini G, Parrini S, Castroflorio T, Deregibus A, Debernardi CL. Efficacy of clear aligners in controlling orthodontic tooth movement: a systematic review. Angle Orthod. 2015 Sep;85(5):881-9. doi: 10.2319/061614-436.1. Epub 2014 Nov 20. PMID 25412265
- [Background] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432
- [Background] Todd MA, Staley RN, Kanellis MJ, Donly KJ, Wefel JS. Effect of a fluoride varnish on demineralization adjacent to orthodontic brackets. Am J Orthod Dentofacial Orthop. 1999 Aug;116(2):159-67. doi: 10.1016/s0889-5406(99)70213-1. PMID 10434089
- [Background] Banks PA, Chadwick SM, Asher-McDade C, Wright JL. Fluoride-releasing elastomerics--a prospective controlled clinical trial. Eur J Orthod. 2000 Aug;22(4):401-7. doi: 10.1093/ejo/22.4.401. PMID 11029829
- [Background] Benson PE, Douglas CW, Martin MV. Fluoridated elastomers: effect on the microbiology of plaque. Am J Orthod Dentofacial Orthop. 2004 Sep;126(3):325-30. doi: 10.1016/j.ajodo.2003.07.007. PMID 15356496
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Gay G, Ravera S, Castroflorio T, Garino F, Rossini G, Parrini S, Cugliari G, Deregibus A. Root resorption during orthodontic treatment with Invisalign(R): a radiometric study. Prog Orthod. 2017 Dec;18(1):12. doi: 10.1186/s40510-017-0166-0. Epub 2017 May 15. PMID 28503724
- [Background] Bisht S, Khera AK, Raghav P. White spot lesions during orthodontic clear aligner therapy: A scoping review. J Orthod Sci. 2022 May 4;11:9. doi: 10.4103/jos.jos_170_21. eCollection 2022. PMID 35754408
- [Background] Sudjalim TR, Woods MG, Manton DJ. Prevention of white spot lesions in orthodontic practice: a contemporary review. Aust Dent J. 2006 Dec;51(4):284-9; quiz 347. doi: 10.1111/j.1834-7819.2006.tb00445.x. PMID 17256301
- [Background] Horst JA, Tanzer JM, Milgrom PM. Fluorides and Other Preventive Strategies for Tooth Decay. Dent Clin North Am. 2018 Apr;62(2):207-234. doi: 10.1016/j.cden.2017.11.003. PMID 29478454
- [Background] Benson PE, Parkin N, Dyer F, Millett DT, Germain P. Fluorides for preventing early tooth decay (demineralised lesions) during fixed brace treatment. Cochrane Database Syst Rev. 2019 Nov 17;2019(11):CD003809. doi: 10.1002/14651858.CD003809.pub4. PMID 31742669
- [Background] Stecksen-Blicks C, Renfors G, Oscarson ND, Bergstrand F, Twetman S. Caries-preventive effectiveness of a fluoride varnish: a randomized controlled trial in adolescents with fixed orthodontic appliances. Caries Res. 2007;41(6):455-9. doi: 10.1159/000107932. Epub 2007 Sep 7. PMID 17827963
- [Background] Sajjan PG, Nagesh L, Sajjanar M, Reddy SK, Venktesh UG. Comparative evaluation of chlorhexidine varnish and fluoride varnish on plaque Streptococcus mutans count--an in vivo study. Int J Dent Hyg. 2013 Aug;11(3):191-7. doi: 10.1111/idh.12028. Epub 2013 May 30. PMID 23721577
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Houston WJ. The analysis of errors in orthodontic measurements. Am J Orthod. 1983 May;83(5):382-90. doi: 10.1016/0002-9416(83)90322-6. PMID 6573846
- [Background] Sonesson M, Brechter A, Abdulraheem S, Lindman R, Twetman S. Fluoride varnish for the prevention of white spot lesions during orthodontic treatment with fixed appliances: a randomized controlled trial. Eur J Orthod. 2020 Jun 23;42(3):326-330. doi: 10.1093/ejo/cjz045. PMID 31197364
- [Background] Restrepo M, Bussaneli DG, Jeremias F, Cordeiro RC, Magalhaes AC, Palomari Spolidorio DM, Santos-Pinto L. Control of white spot lesion adjacent to orthodontic bracket with use of fluoride varnish or chlorhexidine gel. ScientificWorldJournal. 2015;2015:218452. doi: 10.1155/2015/218452. Epub 2015 Apr 20. PMID 25973442
- [Background] Paula AB, Fernandes AR, Coelho AS, Marto CM, Ferreira MM, Caramelo F, do Vale F, Carrilho E. Therapies for White Spot Lesions-A Systematic Review. J Evid Based Dent Pract. 2017 Mar;17(1):23-38. doi: 10.1016/j.jebdp.2016.10.003. Epub 2016 Nov 1. PMID 28259311
- [Background] Azarpazhooh A, Limeback H. Clinical efficacy of casein derivatives: a systematic review of the literature. J Am Dent Assoc. 2008 Jul;139(7):915-24; quiz 994-5. doi: 10.14219/jada.archive.2008.0278. PMID 18594077
- [Background] van Loveren C, Duggal MS. Experts' opinions on the role of diet in caries prevention. Caries Res. 2004;38 Suppl 1:16-23. doi: 10.1159/000074358. PMID 14685020
- [Background] Xie Z, Yu L, Li S, Li J, Liu Y. Comparison of therapies of white spot lesions: a systematic review and network meta-analysis. BMC Oral Health. 2023 Jun 1;23(1):346. doi: 10.1186/s12903-023-03076-x. PMID 37264364
- [Background] Yassir YA, Nabbat SA, McIntyre GT, Bearn DR. Clinical effectiveness of clear aligner treatment compared to fixed appliance treatment: an overview of systematic reviews. Clin Oral Investig. 2022 Mar;26(3):2353-2370. doi: 10.1007/s00784-021-04361-1. Epub 2022 Jan 6. PMID 34993617
- [Background] Raghavan S, Abu Alhaija ES, Duggal MS, Narasimhan S, Al-Maweri SA. White spot lesions, plaque accumulation and salivary caries-associated bacteria in clear aligners compared to fixed orthodontic treatment. A systematic review and meta- analysis. BMC Oral Health. 2023 Aug 27;23(1):599. doi: 10.1186/s12903-023-03257-8. PMID 37635207
- [Background] Al Saffan AD. Current Approaches to Diagnosis of Early Proximal Carious Lesion: A Literature Review. Cureus. 2023 Aug 14;15(8):e43489. doi: 10.7759/cureus.43489. eCollection 2023 Aug. PMID 37719595
- [Background] Al-Khateeb S, Forsberg CM, de Josselin de Jong E, Angmar-Mansson B. A longitudinal laser fluorescence study of white spot lesions in orthodontic patients. Am J Orthod Dentofacial Orthop. 1998 Jun;113(6):595-602. doi: 10.1016/s0889-5406(98)70218-5. PMID 9637561
- [Background] Lucchese A, Gherlone E. Prevalence of white-spot lesions before and during orthodontic treatment with fixed appliances. Eur J Orthod. 2013 Oct;35(5):664-8. doi: 10.1093/ejo/cjs070. Epub 2012 Oct 8. PMID 23045306
- [Background] Sardana D, Ekambaram M, Yang Y, McGrath CP, Yiu CKY. Caries-preventive effectiveness of two different fluoride varnishes: A randomised clinical trial in patients with multi-bracketed fixed orthodontic appliances. Int J Paediatr Dent. 2023 Jan;33(1):50-62. doi: 10.1111/ipd.13013. Epub 2022 Jul 10. PMID 35737872
- [Background] Benson PE, Parkin N, Dyer F, Millett DT, Furness S, Germain P. Fluorides for the prevention of early tooth decay (demineralised white lesions) during fixed brace treatment. Cochrane Database Syst Rev. 2013 Dec 12;(12):CD003809. doi: 10.1002/14651858.CD003809.pub3. PMID 24338792
- [Background] Baik A, Alamoudi N, El-Housseiny A, Altuwirqi A. Fluoride Varnishes for Preventing Occlusal Dental Caries: A Review. Dent J (Basel). 2021 Jun 3;9(6):64. doi: 10.3390/dj9060064. PMID 34204978
- [Background] Quock RL, Warren-Morris DP. Fluoride varnish: the top choice for professionally applied fluoride. Tex Dent J. 2010 Aug;127(8):749-59. PMID 20945734
- [Background] Sonesson M, Twetman S. Prevention of white spot lesions with fluoride varnish during orthodontic treatment with fixed appliances: a systematic review. Eur J Orthod. 2023 Sep 18;45(5):485-490. doi: 10.1093/ejo/cjad013. PMID 37032523
- [Background] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Background] Moshiri M, Eckhart JE, McShane P, German DS. Consequences of poor oral hygiene during aligner therapy. J Clin Orthod. 2013 Aug;47(8):494-8. No abstract available. PMID 24121400